CLINICAL TRIAL: NCT04265703
Title: Central Venous Access in Patients With Difficult Cannulation, A Randomized Controlled Trial
Brief Title: The INVADE Study: INnominate Vein Approach for Central Catheterization in Difficult to cannulatE Patients
Acronym: INVADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Collaborators: Instituto Jalisciense de Cancerologia (Other Government)
Responsible Party: Principal Investigator, Miguel Á Ibarra-Estrada, Principal Investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCG/CEI-1196/19
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness
Keywords: Central venous access; Ultrasound-guided catheterization; Innominate vein; Brachiocephalic vein
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Internal jugular vein site (Active Comparator): Ultrasound-guided central venous catheterization at internal jugular vein site
  Interventions: Procedure: Internal jugular vein catheterization
- Subclavian vein site (Active Comparator): Ultrasound-guided central venous catheterization at subclavian vein site
  Interventions: Procedure: Subclavian vein catheterization
- Innominate vein site (Active Comparator): Ultrasound-guided central venous catheterization at innominate vein site
  Interventions: Procedure: Innominate vein catheterization

INTERVENTIONS:
Procedure: Internal jugular vein catheterization — Catheterization of internal jugular vein with real-time (in-plane) method, with neutral neck position. Standard aseptic technique.
  Arms: Internal jugular vein site
Procedure: Subclavian vein catheterization — Catheterization of subclavian/axillary vein with infra-clavicular approach with real-time (in-plane) method, without shoulder retraction. Standard aseptic technique.
  Arms: Subclavian vein site
Procedure: Innominate vein catheterization — Catheterization of innominate vein with supra-clavicular approach with real-time (in-plane) method, with neutral shoulder position and no shoulder retraction. Standard aseptic technique.
  Arms: Innominate vein site

SUMMARY:
Most recent guidelines suggest central venous access must be performed with real-time ultrasound guidance, and the most recommended site for cannulation is internal jugular vein (IJV); however, it is recognized that evidence for other sites is, at present, limited. Besides, guidelines does not account for patients with small vein cross-sectional area and/or respirophasic collapse, which can make the procedure more difficult or even impossible. The investigators aim to compare three different insertion sites for central venous access, with real-time ultrasound guidance

DETAILED DESCRIPTION:
Ultrasound-guided cannulation of central veins is successful in >95% of the cases, according to the largest study so far. However, this and other studies with similar success rate, are performed in patients with general anesthesia and/or neuromuscular blockade, without spontaneous respiratory efforts. Critical care physicians and many other specialists frequently need to cannulate patients in special circumstances as hypovolemia, pain, anxiety, and respiratory efforts that promotes respirophasic variation in cross-sectional area, and even complete collapse of the vessel. These changes can increase the probability of posterior wall or arterial puncture, hematomas, pneumothorax, etc. Supraclavicular approach for cannulation of the subclavian vein is a method described since 1965, also giving direct access to the innominate vein, a larger vessel which is rarely collapsible regardless of volume status or respiratory efforts. Based on a previous pilot trial, in this multi-center, prospective, randomized, controlled trial, the investigators aim to compare the successfulness and safety of ultrasound-guided central venous cannulation at 3 different sites: internal jugular, subclavian, and innominate veins.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need central venous catheterization, and have respirophasic variation in cross-sectional area of jugular veins

Exclusion Criteria:

* Less than 18 years-old

  * Patients with previous failed attempts with non-ultrasound guided technique
  * Non-resolved pneumothorax/hemothorax at enrollment
  * Refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Cannulation failure rate | Baseline
  Failure to cannulate selected vein at first attempt

SECONDARY OUTCOMES:
Central line-associated blood infection rate | 28 days
  Confirmed with blood cultures
Collapsibility associated with failure | Baseline
  Percentage of vein collapsibility independently associated with cannulation failure
Cannulation number of attempts | Baseline
  Number of attempts needed to attain cannulation
Procedure time | Baseline
  Time from skin puncture to guidewire confirmed into vessel (minutes)
Arterial puncture rate | Baseline
  Confirmed immediately after procedure with vascular ultrasound
Hematoma formation rate | 7 days
  Confirmed immediately after procedure with vascular ultrasound
Neumothorax rate | 7 days
  Confirmed immediately after procedure with lung ultrasound
Hemothorax rate | 7 days
  Confirmed immediately after procedure with lung ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ibarra-Estrada, MD, Principal Investigator — Hospital Civil Fray Antonio Alcalde
Locations (1):
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: No